CLINICAL TRIAL: NCT03528993
Title: The Effect of Exercise by Mechanical Hippotherapy Device on Postural Stability and Balance in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, osman coban, PT, MSc, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-02
Record Dates: First submitted 2018-04-23; First posted 2018-05-18 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Stroke; Gait, Hemiplegic; Balance, Postural
Keywords: stroke, hippotherapy, balance, postural control, gait
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise by hippotherapy device group (Experimental): The experimental group receive conventional rehabilitation for 45 min/day following by use of a hippotherapy device for 15 min/day, 5 times/week for 4 weeks
  Interventions: Other: exercise by hippotherapy device; Other: conventional rehabilitation
- Control group (Other): The control group will receive conventional rehabilitation for 45 min/day, following by postural control exercises 15 min/day 5 times/week for 4 weeks.
  Interventions: Other: conventional rehabilitation; Other: postural control exercises

INTERVENTIONS:
Other: exercise by hippotherapy device — Hippotherapy device mostly used on cerebral palsy, but we want to use hippotherapy device on patient with Hemiplegia.
  Arms: Exercise by hippotherapy device group
Other: conventional rehabilitation — Bobath exercises: Bobath is a type of physiotherapy treatment which aims to improve movement and mobility in patients with damage to their central nervous system (brain and spinal cord).
Other: postural control exercises — perturbation on four directions, weight bearing exercises on standing positions
  Arms: Control group

SUMMARY:
Stroke,one of the leading cause of death, is caused by ischemia or hemorrhage. It results in neurological deficits such as hemiplegia. Hemiplegia show disability characterized loss of motor, sensory and cognitive function. Reduced postural control and balance stability results gait disturbances such as asymmetric weight bearing, risk of falling and imbalances. It also shows increased energy expenditure, decreased independence on quality of life and limited mobility. Physical therapy can be effective method for solving these problems. Hippotherapy, also known as horseback riding therapy, is a form of physical therapy strategy that uses equine movement. The concept of hippotherapy is to use a horse as a therapeutic tool, and it is based on similarities in gait between the human and horse. The horse's gait provides patients having motor disabilities with rhythmic and repetitive movements similar to human walking, thereby giving them training opportunities to improve posture, balance, and strength. Even though it has many effect on solving these problems, hippotherapy centers are not enough. Due to climate and environmental situations, hippotherapy devices were improved and had similar effects on patients with stroke. In literature, these device mostly used on cerebral palsy, but investigator wants to use hippotherapy device on patient with Hemiplegia. For these reasons, the effects of exercises by mechanical hippotherapy device on postural control and balance will be investigated.

DETAILED DESCRIPTION:
Investigator will randomly allocate 30 patients with hemiplegia to two groups; Control group (n=15), experimental group(n=15).The control group will receive conventional rehabilitation for 45 min/day, following by postural control exercises 15 min/day 5 times/week for 4 weeks, while the experimental group receive conventional rehabilitation for 45 min/day following by use of a hippotherapy device for 15 min/day, 5 times/week for 4 weeks. Assessment procedure will be held at the beginning and 4th week of study. Assessment procedure will be held at the beginning and 4th week of study. All subjects will be assessed by berg balance scale and BIODEX primarily while Timed up and go test, SF-36, Functional reach test, functional independence measurement(FIM), Trunk Impairment Scale (TIS), Trunk Control Test (TCT), motricity index, Fugl-meyer will be held secondarily.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental Test score more than 24
* Ability to stand and sit independently
* Ability to follow and understand verbal instructions.

Exclusion criteria:

* Musculoskeletal problems
* Neurologic deficits such as unilateral neglect, hemianopsia, and apraxia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | Change from baseline to week 4
  The Berg Balance Scale (BBS) was developed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks. It is a valid instrument used for evaluation of the effectiveness of interventions and for quantitative descriptions of function in clinical practice and research. The BBS has been evaluated in several reliability studies. A recent study of the BBS, which was completed in Finland, indicates that a change of eight (8) BBS points is required to reveal a genuine change in function between two assessments among older people who are dependent in ADL and living in residential care facilities. 14-item scale designed to measure balance of the older adult in a clinical setting. Equipment needed: Ruler, two standard chairs (one with arm rests, one without), footstool or step, stopwatch or wristwatch, 15 ft walkway Completion Time: 15-20 minutes
BIODEX balance systems | Change from baseline to week 4
  Biodex Balance System (BBS), a commercially available balance device, Biodex Medical Systems, Shirley, NY, USA) will used to assess fall risk and balance. It consists of a movable balance platform which provides up to 20° of surface tilt in a 360° range of motion and the platform is interfaced with computer software (Upper display module-firmware version 1.09, Lower control board-firmware version 1.03, Biodex Medical Systems) that enables the device to serve as an objective assessment of balance and fall risk. The system had various difficulty levels which range from 1 (most difficult) to 12 (the easiest). two settings will be used to assess the dynamic balance and the fall risk;the postural stability test (PST) and the fall risk test (FRT).

SECONDARY OUTCOMES:
Timed Up and Go Test | Change from baseline to week 4
  This test was initially designed for elderly persons To determine fall risk and measure the progress of balance, sit to stand, and walking, is used for people with stroke, Parkinsons, Multiple Sclerosis, hip fracture, Alzheimer, Huntington Disease and others.
SF-36 (The Short Form Health Survey) | Change from baseline to week 4
  The Short Form-36 (SF-36) is a 36 item questionnaire which measures Quality of Life (QoL) across eight domains, which are both physically and emotionally based. The eight domains that the SF36 measures are as follows: physical functioning; role limitations due to physical health; role limitations due to emotional problems; energy/fatigue; emotional well-being; social functioning; pain; general health. A single item is also included that identifies perceived change in health, making the SF-36 a useful indicator for change in QoL over time and treatment.
Functional Reach Test | Change from baseline to week 4
  The Functional Reach Test was first developed by Pamela Duncan and colleagues in 1990. It is a quick and simple, single-task dynamic test that defines functional reach as "the maximal distance one can reach forward beyond arm's length, while maintaining a fixed base of support in the standing position". It is a dynamic rather than a static test and measures a person's "margin of stability" as well as ability to maintain balance during a functional task. The test has been shown by Duncan to be predictive of falls in older adults.
Functional Independence Measurement(FIM) | Change from baseline to week 4
  The Functional Independence Measure (FIM) is an 18-item of physical, psychological and social function. The tool is used to assess a patient's level of disability as well as change in patient status in response to rehabilitation or medical intervention. Tasks that are evaluated using the FIM include bowel and bladder control, transfers, locomotion, communication, social cognition as well as the following six self-care activities: Feeding,Grooming, Bathing, Upper Body Dressing, Lower Body Dressing,Toileting
Fugl-Meyer Assessment of Motor Recovery after Stroke | Change from baseline to week 4
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. The scale is comprised of five domains and there are 155 items in total: Motor functioning (in the upper and lower extremities), Sensory functioning (evaluates light touch on two surfaces of the arm and leg, and position sense for 8 joints), Balance (contains 7 tests, 3 seated and 4 standing), Joint range of motion (8 joints), Joint pain.
The Trunk Control Test (TCT) | Change from baseline to week 4
  The Trunk Control Test can be used to assess the motor impairment in a patient who has had a stroke. It correlates with eventual walking ability. It has 4 items: 1) Rolling to weak side 2) Rolling to strong side 3) Balance in sitting position 4) Sit up from lying down. Total score range: 0 (minimum) to 100 (maximum, indicating better performance). Score of each item: (0, 12 or 25). 0 = unable to perform movement without assistance. 12 = able to perform movement, but in an abnormal style 25 = able to complete movement normally. For the sitting balance item, a patient scores 12 if they need to touch anything with their hands to stay upright, and 0 if they are unable to stay up (by any means) for 30 seconds.
Trunk Impairment Scale (TIS) | Change from baseline to week 4
  Trunk Impairment Scale (TIS) measures the motor impairment of the trunk after a stroke through the evaluation of static and dynamic sitting balance as well as co-ordination of trunk movement. The static subscale investigates: (1) the ability of the subject to maintain a sitting position; (2) the ability to maintain a sitting position while the legs are passively crossed, (3) the ability to maintain a sitting position when the subject crosses the legs actively. The dynamic subscale contains items on L. flexion of the trunk and unilateral lifting of the hip. To assess the coordination of the trunk, the subject is asked to rotate the upper or lower part of his or her trunk 6 times, Scores range from a minimum of 0 to a maximum of 23. If patient scores 0 on the first item, the total score on the TIS is 0.

CONTACTS AND LOCATIONS:
Overall Officials: fatma mutluay, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee CW, Kim SG, Yong MS. Effects of hippotherapy on recovery of gait and balance ability in patients with stroke. J Phys Ther Sci. 2014 Feb;26(2):309-11. doi: 10.1589/jpts.26.309. Epub 2014 Feb 28. PMID 24648655
- [Background] Han JY, Kim JM, Kim SK, Chung JS, Lee HC, Lim JK, Lee J, Park KY. Therapeutic effects of mechanical horseback riding on gait and balance ability in stroke patients. Ann Rehabil Med. 2012 Dec;36(6):762-9. doi: 10.5535/arm.2012.36.6.762. Epub 2012 Dec 28. PMID 23342307
- [Background] Sung YH, Kim CJ, Yu BK, Kim KM. A hippotherapy simulator is effective to shift weight bearing toward the affected side during gait in patients with stroke. NeuroRehabilitation. 2013;33(3):407-12. doi: 10.3233/NRE-130971. PMID 23949070
- [Derived] Coban O, Mutluay F. The effects of mechanical hippotherapy riding on postural control, balance, and quality of life (QoL) in patients with stroke. Disabil Rehabil. 2024 Jun;46(11):2338-2347. doi: 10.1080/09638288.2023.2221458. Epub 2023 Jun 11. PMID 37303153